CLINICAL TRIAL: NCT01077752
Title: Effect of Local Anesthetic Continuous Preperitoneal Wound Infiltration on Incisional Hyperalgesia Following Colorectal Laparoscopic Surgery
Brief Title: Local Anesthetic Continuous Preperitoneal Infiltration and Wound Hyperalgesia
Acronym: CATCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AOR 08028
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Pain, Postoperative
Keywords: Pain, postoperative; Local infiltration; Hyperalgesia, postoperative; Local anesthetic, ropivacaine, lidocaine; Colorectal laparoscopic surgery; Pain management after colorectal laparoscopic surgery
MeSH Terms: conditions — Pain, Postoperative; Hyperalgesia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Patients with continuous ropivacaine preperitoneal infusion
  Interventions: Drug: continuous ropivacaine preperitoneal infusion; Drug: parenteral analgesia combining acetaminophen and morphine
- 2 (Active Comparator): Patients with intravenous lidocaine infusion
  Interventions: Drug: intravenous lidocaine infusion; Drug: parenteral analgesia combining acetaminophen and morphine
- 3 (Placebo Comparator): Patients without local anesthetics
  Interventions: Drug: parenteral analgesia combining acetaminophen and morphine; Drug: NaCl

INTERVENTIONS:
Drug: continuous ropivacaine preperitoneal infusion — Bolus of 20 mg after the surgery then 20 mg per hour during 48 hours
  Arms: 1
Drug: intravenous lidocaine infusion — Bolus of 60 mg after the surgery then 60 mg per hour during 48 hours
  Arms: 2
Drug: parenteral analgesia combining acetaminophen and morphine — parenteral analgesia combining acetaminophen and morphine
Drug: NaCl — NaCl
  Arms: 3

SUMMARY:
In this multicenter, randomised, placebo-controlled, double-blind trial, hyperalgesia area around the scarce following colorectal laparoscopic surgery (piece removal) will be assessed in 3 groups of patients : group 1: continuous ropivacaine preperitoneal infusion, group 2 : intravenous lidocaine infusion, or group 3 : control group without local anesthetics. All patients will receive parenteral analgesia combining acetaminophen and morphine.

DETAILED DESCRIPTION:
Besides hyperalgesia assessment, immediate postoperative and long-term pain, morphine consumption, and endocrin-metabolic response will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* ASA status 1 - 3
* Colorectal laparoscopic surgery with piece removal
* French speaking
* Written informed consent

Exclusion Criteria:

* laparoscopy without colorectal extraction
* chronic pain
* analgesic consumption during the 24 hours previous to the surgery
* morphine and LA intolerance
* drug addiction
* inflammatory bowel disease
* general inflammatory disease
* sepsis
* anemia < 10 gr/dl
* liver or renal or cardiac insufficiency
* uncontrolled diabetes
* preoperative consumption of opiate/corticosteroid/beta-blockers, and anti-arrhythmic drugs, MAOIs, neuroleptics.
* preoperative consumption of NSAIDs excluding aspirin referred cardiology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pericicatricial hyperalgesia area | 72 hours after surgery

SECONDARY OUTCOMES:
Pain intensity (rest/mobilization and long-term) | 72 hours, 3 months and 6 months after surgery
Morphine consumption | During 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc Beaussier, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Departement d'Anesthesie-Reanimation, Hopital Saint-Antoine, Paris, France